CLINICAL TRIAL: NCT02161991
Title: Randomized Phase 3 Study of Aprepitant Versus Placebo in Chinese Advanced Non-small Cell Lung Cancer Who Received Highly Emetogenic Chemotherapy
Brief Title: Aprepitant for Chemotherapy Induced Nausea and Vomiting in Chinese Advanced Non-small Cell Lung Cancers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director of department of medical oncology, lung cancer and gastrointestinal cancer unit, Hunan Province Tumor Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACINV
Record Dates: First submitted 2014-06-02; First posted 2014-06-12 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma, Non-small Cell Lung
Keywords: aprepitant; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aprepitant group (Experimental): Patients assigned to aprepitant group should receive aprepitant for the control of CINV, aprepitant 125 mg for day1, 80mg for day2 and day3.
  Interventions: Drug: Aprepitant
- placebo (Placebo Comparator): Patients assigned to placebo group should receive placebo for the control of CINV compared with aprepitant group.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aprepitant — aprepitant should be give when patients receive platinum based chemotherapy, 125mg for day1, 80mg for day2 and day3.
  Other Names: Emend
  Arms: aprepitant group
Drug: placebo — placebo should be give when patients receive platinum based chemotherapy, 125mg for day1, 80mg for day2 and day3.
  Arms: placebo

SUMMARY:
Aprepitant is an oral neurokinin-1(NK-1) antagonist which is widely used for the prevention of chemotherapy-induced nausea and vomiting(CINV), it is metabolized by CYP34A, however, up to now it was still unknown the CINV control rate of aprepitant in Chinese non-small cell lung cancer(NSCLC) patients, we hypothesis that CYP3A4 and NK-1 polymorphism would influence aprepitant plasma concentration, which may lead to the individual difference of CINV control rate.

DETAILED DESCRIPTION:
Patients pathologic diagnosed of advanced non-small cell lung cancer, according to NCCN non-small cell lung cancer guide line(2014 V2),the patient should receive standard platinum based chemotherapy, are randomized divided into two groups, aprepitant group and placebo group. In aprepitant group, patients would receive aprepitant 125 mg at day1, then 80 mg at day2 and day3. In placebo group, patients would receive placebo from day1 to day3. In both group, dexamethasone and 5-HT inhibitor palonosetron were give at the same dose. During the treatment, any grade of nausea and vomiting should be recorded in order to evaluate the complete response rate of CINV, other side-effects should be recorded. In aprepitant group, plasma should be taken for the analyze of plasma concentration, gene polymorphism of CYP3A4 and NK-1 should be analyzed for all the patients who received aprepitant if possible.

ELIGIBILITY:
Inclusion Criteria:

* patients pathologic diagnosed of advanced non-small cell lung cancer
* according to NCCN non-small cell lung cancer guide line(2014 V2), patients are suitable for platinum based chemotherapy.

Exclusion Criteria:

* patients could not receive platinum based chemotherapy judged by clinical doctors
* pregnancy or breast-feeding women
* any serious disease which could not be controled
* urine protein≥++, or 24h urine protein>1g
* less than 18 years old or more than 75 years old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
complete response rate of CINV | during treatment, up to 6 months
  complete response rate of CINV should be recorded when platinum based chemotherapy begun, during inhospital treatment, up to 6 months

SECONDARY OUTCOMES:
adverse event | during treatment, up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

REFERENCES:
- [Background] Hu Z, Cheng Y, Zhang H, Zhou C, Han B, Zhang Y, Huang C, Chang J, Song X, Liang J, Liang H, Bai C, Yu S, Chen J, Wang J, Pan H, Chitkara DK, Hille DA, Zhang L. Aprepitant triple therapy for the prevention of chemotherapy-induced nausea and vomiting following high-dose cisplatin in Chinese patients: a randomized, double-blind, placebo-controlled phase III trial. Support Care Cancer. 2014 Apr;22(4):979-87. doi: 10.1007/s00520-013-2043-9. Epub 2013 Nov 26. PMID 24276953
- [Background] Aapro MS, Schmoll HJ, Jahn F, Carides AD, Webb RT. Review of the efficacy of aprepitant for the prevention of chemotherapy-induced nausea and vomiting in a range of tumor types. Cancer Treat Rev. 2013 Feb;39(1):113-7. doi: 10.1016/j.ctrv.2012.09.002. Epub 2012 Oct 11. PMID 23062719
- [Background] Stiff PJ, Fox-Geiman MP, Kiley K, Rychlik K, Parthasarathy M, Fletcher-Gonzalez D, Porter N, Go A, Smith SE, Rodriguez TE. Prevention of nausea and vomiting associated with stem cell transplant: results of a prospective, randomized trial of aprepitant used with highly emetogenic preparative regimens. Biol Blood Marrow Transplant. 2013 Jan;19(1):49-55.e1. doi: 10.1016/j.bbmt.2012.07.019. Epub 2012 Aug 1. PMID 22863840
- [Background] Albany C, Brames MJ, Fausel C, Johnson CS, Picus J, Einhorn LH. Randomized, double-blind, placebo-controlled, phase III cross-over study evaluating the oral neurokinin-1 antagonist aprepitant in combination with a 5HT3 receptor antagonist and dexamethasone in patients with germ cell tumors receiving 5-day cisplatin combination chemotherapy regimens: a hoosier oncology group study. J Clin Oncol. 2012 Nov 10;30(32):3998-4003. doi: 10.1200/JCO.2011.39.5558. Epub 2012 Aug 20. PMID 22915652